CLINICAL TRIAL: NCT04612920
Title: Towards Enhanced Recovery After Cesarean: Scheduled Post-operative Medication: a Randomized Controlled Trial
Brief Title: Towards Enhanced Recovery After Cesarean
Acronym: ERAS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 12675
Record Dates: First submitted 2020-10-15; First posted 2020-11-03 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Cesarean Section Complications
MeSH Terms: interventions — Ibuprofen; Acetaminophen; Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study Group (Experimental): Participants will receive ibuprofen 800mg every eight hours and acetaminophen 1000mg every eight hours, given at the same time, along with oxycodone five mg every six hours PRN for breakthrough pain.
  Interventions: Drug: Ibuprofen, acetaminophen, oxycodone
- Standard Group (No Intervention): Participants will receive current OU standard of care therapy which includes ibuprofen 800mg every eight hours as needed (PRN), acetaminophen 1000mg every eight hours PRN, and oxycodone five mg every six hours PRN.

INTERVENTIONS:
Drug: Ibuprofen, acetaminophen, oxycodone — The timing of medications is the intervention.
  Arms: Study Group

SUMMARY:
One in 300 women will become persistent opioid users after cesarean delivery (1). Cesarean delivery is the most common surgical procedure in the United States, representing 31.9% of the 3,788,235 deliveries in 2018 (2). Patients have to cope with the pain and challenges of post-operative care while adjusting to motherhood and completing activities of daily living. Often when they return home, they are also tasked with other domestic roles which compounds the challenge of this post-operative period. With a potential impact just in the US on 1.2 million mothers each year, optimizing post-operative pain management in order to reduce the risk of persistent opioid use represents an urgent unmet public health goal. To this end, there are national efforts to reduce the cesarean rate and optimize post-cesarean pain management (3,4). The majority of efforts in the last few years have focused on home-going medications and alterations in prescription practices. Recent recommendations from the Enhanced Recovery After Surgery Society indicate that patients should receive multi-modal analgesia on a regular basis, along with early post-delivery mobilization (3). However, the efficacy of scheduled non-steroidal anti-inflammatory medications (NSAID) along with acetaminophen in the immediate post-operative period and after going home have not been systematically studied in the cesarean population. We hypothesize that patients who receive scheduled medications in the post-operative period are less likely to require opioids for pain relief both in the hospital and after they return home.

DETAILED DESCRIPTION:
The proposed study is a pragmatic randomized control trial of post-cesarean pain management techniques with participants allocated in a 1:1 ratio using a random block allocation table using blocks of size 4 and 6. Given the nature of the study, it would be impossible to blind participants and clinicians. Participants will be randomized after completion of the procedure to ensure that patients who have significant surgical complications such as severe hemorrhage or those undergoing hysterectomy are excluded.

All participants will receive intrathecal morphine 150mcg per OU standard of care, with orders for pain management per anesthesia for the first 24 hours with a regular diet, removal of urinary catheter 12-24 hours post-operatively, and abdominal binder placed after surgery. In addition, patients will be provided with a fitness tracker to be worn on their wrist throughout hospitalization and until their post-operative visit. After 24 hours, participants will be assigned to either receive current OU standard of care therapy which includes ibuprofen 800mg every eight hours as needed (PRN), acetaminophen 1000mg every eight hours PRN, and oxycodone five mg every six hours PRN or the study protocol. The study protocol will include scheduled ibuprofen 800mg every eight hours and acetaminophen 1000mg every eight hours, given at the same time, along with oxycodone five mg every six hours PRN for breakthrough pain. Both sets of patients will be provided with 60 pills of acetaminophen 500mg and 30 pills ibuprofen 800mg to take at home, with the study participants receiving instructions to take the medications in a scheduled fashion and the other group in an as needed fashion. Both groups will receive a discharge prescription for 20 pills of oxycodone five mg every 6 hours PRN to be taken for breakthrough pain as needed--current standard at OU. All prescriptions will be delivered to the patient from the pharmacy prior to discharge per our departmental standard. Patient requiring more medications to control pain beyond the randomized approach described above will be treated per the discretion of the attending physician or designee. Patients will be seen for a post-operative care visit on post discharge day 8-12 depending on patient and clinic availability and asked to bring their fitness tracker and medication bottles with them for assessment of steps taken, medication consumed, pain outcomes and satisfaction scores. The Oklahoma PMP Aware system will be accessed to record prescriptions for controlled substances from other providers.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing repeat cesarean delivery
* ≥37 week gestation
* attended at least 7 prenatal visits
* age ≥18.

Exclusion Criteria:

* Non-English speaking, attended < 7 prenatal visits, fetal anomalies or death, inability to ambulate, BMI ≥45kg/m2 at delivery due to higher risk of regional analgesia complications, placental implantation abnormalities, maternal diabetes due to the risk of wound complications, chorioamnionitis, allergy to study medications, underlying renal or hepatic impairment, opioid use in the last 3 months, chronic controlled substance use, chronic pain disorders, history of narcotic addiction, intraoperative hemorrhage not controlled with medication alone, additional concurrent surgeries other than sterilization procedures and presence of endometriosis noted at time of surgery. Patients will be enrolled and randomized to their respective groups after completion of the surgery, as there may be surgical complications that preclude their final enrollment as described in the exclusion criteria.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only females undergoing cesarean section are eligible.
Enrollment: 33 (Actual)
Dates: Start 2020-12-12 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Amount of morphine milligram equivalents used from 25-72 hours post-op | 25-72 hours post-op
  Patient's inpatient chart will be reviewed to calculate the amount of oxycodone the patient used, converted to morphine milligram equivalents and recorded.
Patient's morphine milligram equivalent usage from day of discharge to outpatient post-operative visit | post-discharge day #8-12
  The patient will be discharged home with 20 tablets of oxycodone 5mg. When they return to their post-operative visit, we will count the number of tablets left in the pill bottle. A low number of remaining tablets would mean increased medication usage outpatient.

SECONDARY OUTCOMES:
Patient's pain rating on post-operative day #2 and #3 with and without ambulation | post-op days #2 and #3
  The patient will be asked to rate her pain on post-operative day #2 and #3 with and without ambulation on a scale from 1-10 with 1 representing severe pain and 10 representing well controlled pain.
Patient's pain satisfaction scale on day of post-operative visit | 1 day of post-operative visit
  Patient will be asked to mark on a line how satisfied she is with her pain management outpatient with the left side of the line representing poor satisfaction and the right side of the line representing good satisfaction with pain control. The place she marks on the line will be measured and recorded in centimeters.
Patient's pain satisfaction scale on day of discharge | 1 day of discharge
  Patient will be asked to mark on a line how satisfied she is with her pain management during admission with the left side of the line representing poor satisfaction and the right side of the line representing good satisfaction with pain control. The place she marks on the line will be measured and recorded in centimeters.
Amount of acetaminophen used on post-operative day #2 and #3 | post-operative day #2 and #3
  Chart will be reviewed to calculate the amount of acetaminophen in milligrams the patient required on post-operative day #2 and #3 from 0000 to 2359.
Amount of ibuprofen used on post-operative day #2 and #3 | post-operative days #2 and #3
  Chart will be reviewed to calculate the amount of ibuprofen in milligrams the patient required on post-operative day #2 and #3 from 0000 to 2359.
Amount a patient ambulates on post-operative day #2 and #3 | post-operative day #2 and #3
  The patient will be given a fitness tracker after surgery and the number of steps the patient takes on post-operative day #2 and #3 will be recorded from 0000 to 2359.
Patient's readiness to be discharged | post-operative day #2 and #3
  A validated questionnaire will be administered on post-operative day #2 and #3 by a research nurse assessing the patient's perceived readiness to be discharged home.
Patient's ambulation on outpatient day #1-3 | information from outpatient day #1-3 will be recorded at the patient's post-operative visit
  The patient will be given a fitness tracker after surgery and the number of steps the patient takes on outpatient day #1-3 will be recorded daily from 0000 to 2359.
Patient's ambulation on outpatient day #4-5 | information from outpatient day #4-5 will be recorded at the patient's post-operative visit
  The patient will be given a fitness tracker after surgery and the number of steps the patient takes on outpatient day #4-5 will be recorded daily from 0000 to 2359.
Patient's sleep pattern on outpatient night #1-3 | information from outpatient night #1-3 will be recorded at the patient's post-operative
  The patient will be given a fitness tracker and asked to wear it while sleeping. The amount of time spent in deep sleep, light sleep, and awake will be recorded in hours and minutes on outpatient night #1-3.
Patient's sleep pattern on outpatient night #4-5 | information from outpatient night #4-5 will be recorded at the patient's post-operative visit
  The patient will be given a fitness tracker and asked to wear it while sleeping. The amount of time spent in deep sleep, light sleep, and awake will be recorded in hours and minutes on outpatient night #4-5.
Patient's acetaminophen usage from discharge to outpatient post-operative visit | information will be collected at the outpatient post-operative 1 day visit
  The patient will be discharged home with acetaminophen 500mg. When they return to their post-operative visit, we will count the number of tablets left in the pill bottle. A low number of remaining tablets would mean increased medication usage outpatient.
Patient's ibuprofen usage from discharge to outpatient post-operative visit | information will be collected at the outpatient post-operative 1 day visit
  The patient will be discharged home with ibuprofen 800mg. When they return to their post-operative visit, we will count the number of tablets left in the pill bottle. A low number of remaining tablets would mean increased medication usage outpatient.
Patient's pain rating on day of post-operative visit with and without ambulation | 1 day of post-operative visit
  The patient will be asked to rate her pain at post-operative day with and without ambulation on a scale from 1-10 with 1 representing severe pain and 10 representing well controlled pain.
Patient's pain rating at 12 hours post-op | 12 hours post-op
  The patient will be asked to rate her pain at 12 hour post-op on a scale from 1-10 with 1 representing severe pain and 10 representing well controlled pain.

CONTACTS AND LOCATIONS:
Overall Officials: Pavan Parikh, MD, Principal Investigator — University of Oklahoma HSC
Locations (1):
- University ofOklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No